CLINICAL TRIAL: NCT06613347
Title: Clinical Study to Assess the Efficacy of Professional Tooth Whitening Maintenance System of a Colgate Regimen
Brief Title: Clinical Study to Assess the Efficacy of Professional Tooth Whitening Maintenance System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CRO-2024-07-WHT- SPMW-BGS_ MH
Record Dates: First submitted 2024-09-20; First posted 2024-09-25 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Staining
Keywords: whitening; stains; perceptions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Whitening Regimen (Experimental)
  Interventions: Other: whitening maintenance
- Whitening MW (Active Comparator)
  Interventions: Other: whitening maintenance MW
- Negative Control (Placebo Comparator)
  Interventions: Other: negative control

INTERVENTIONS:
Other: whitening maintenance — whitening maintenance regimen
  Other Names: whitening maintenance regimen
  Arms: Whitening Regimen
Other: whitening maintenance MW — maintenance MW
  Arms: Whitening MW
Other: negative control — negative control
  Arms: Negative Control

SUMMARY:
Clinical study to assess the efficacy of professional tooth whitening maintenance system of a Colgate toothpaste containing 5% Hydrogen Peroxide with a stain-fighter mouthwash as compared to only the stainfighter mouthwash and a negative control toothpaste

ELIGIBILITY:
Inclusion Criteria:

* permanent natural teeth (6-11) (22-27)
* composite lobene =>1
* Signed Informed Consent Form
* Male and female subjects aged 18-70 years, inclusive
* Good general health and good oral health based on the opinion of the study investigator
* All maxillary anterior teeth (teeth #6 through #11) must be present;& mandibular anterior ( Teeth #22 through 27) must be present
* Availability for the duration of the study
* Minimum average Vita Extended Bleachedguide 3D-Master shade score of 17 ≥ or darker
* A minimum mean of 1.5 ≥ determined by the Interproximal Modified Lobene (IML) Stain Index
* Demonstrate a tendency to form stain in anterior teeth/ Have high staining habits ( coffee/ wine/ tea drinker)

Exclusion Criteria:

* allergies
* Presence of orthodontic appliances or any anterior tooth with a prosthetic crown or veneer
* Restorations on the tooth to be scored which may interfere with scoring procedures
* Obvious signs of periodontal disease, rampant caries, or any condition that the dental examiner considers exclusionary from the study
* Five or more carious lesions requiring immediate care
* Concurrent participation in another clinical study
* Self-reported pregnant and/or lactating women
* History of allergies to tooth whitening products, hydrogen peroxide, personal care consumer products, or their ingredients
* Have dentinal sensitivity
* Taking medication within a year which could alters natural tooth color or appearance,
* Have used Professional Whitening product within a year or had a dental prophylaxis ( professional dental cleaning) within 30 days prior to the start of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Tooth color assessment | Baseline
  Changes in Tooth color determined by examiner use of Vita Extended Bleachedguide 3D-Master®(29 tabs)
Tooth color assessment | 4 weeks
  Changes in Tooth color determined by examiner use of Vita Extended Bleachedguide 3D-Master®(29 tabs)
Tooth color assessment | 8 weeks
  Changes in Tooth color determined by examiner use of Vita Extended Bleachedguide 3D-Master®(29 tabs)
Interproximal Modified Lobene Stain Index | Baseline
  Stain examination will be determined by the Interproximal Modified Lobene(IML) Stain Index
Interproximal Modified Lobene Stain Index | 4 week
  Stain examination will be determined by the Interproximal Modified Lobene(IML) Stain Index
Interproximal Modified Lobene Stain Index | 8 week
  Stain examination will be determined by the Interproximal Modified Lobene(IML) Stain Index

CONTACTS AND LOCATIONS:
Locations (1):
- FAR Oral and Systemic Health Consulting, Inc, Costa Mesa, California, United States

IPD SHARING:
Plan to Share IPD: No
It will report only results as aggregate